CLINICAL TRIAL: NCT02157584
Title: A Phase 1, Randomized, Single Center, Open Label, 2 Sequence, 2 Period, Crossover Study to Evaluate the Effect of Food on the Single Dose Pharmacokinetics of Telotristat Etiprate (LX1606 Hippurate) in Healthy Male and Female Subjects
Brief Title: An Open-Label Food Effect Study of Telotristat Etiprate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-107-NRM; LX1606.107 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — telotristat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Subjects will receive a single 500 mg (as free base) dose of telotristat etiprate (as 2 × 250 mg tablets) on Day 1 in a fed condition. Days 2 to 5 will be Washout Days. On Day 6, subjects will receive a single 500 mg (as free base) dose of telotristat etiprate (as 2 × 250 mg tablets) 1 in a fasted condition.
  Interventions: Drug: Telotristat etiprate
- Treatment B (Experimental): Subjects will receive a single 500 mg (as free base) dose of telotristat etiprate (as 2 × 250 mg tablets) on Day 1 in a fasted condition. Days 2 to 5 will be Washout Days. On Day 6, subjects will receive a single 500 mg (as free base) dose of telotristat etiprate (as 2 × 250 mg tablets) 1 in a fed condition.
  Interventions: Drug: Telotristat etiprate

INTERVENTIONS:
Drug: Telotristat etiprate — 2 × 250 mg (as free base) telotristat etiprate tablets (fed conditions /high-fat / high caloric meal)
  Arms: Treatment A
Drug: Telotristat etiprate — 2 × 250 mg (as free base) telotristat etiprate tablets (fasted conditions)
  Arms: Treatment B

SUMMARY:
This study is designed to evaluate the effect of food on the pharmacokinetics (PK) of telotristat ethyl and its metabolite LP-778902 relative to administration of single dose telotristat etiprate in the fasted state in healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects aged ≥18 to ≤55 years of age at screening
* Body mass index ≥18.0 to ≤32.0 kg/m^2
* Acceptable vital signs at Screening: Systolic blood pressure = 90-140 mm Hg, Diastolic blood pressure = 50-90 mm Hg, Heart rate = 40-100 beats per minute
* Able and willing to ingest an entire high fat/high caloric breakfast meal within 30 minutes
* Willingness to adhere to the restrictions outlined in the protocol
* Able to comprehend and sign the Informed Consent Form

Exclusion Criteria:

* Presence of any clinically significant physical, laboratory, or ECG finding that may interfere with the study in the opinion of the Investigator
* Use of any medications, herbal tea, energy drink, herbal products, or supplements within 14 days of study start
* Receipt of any investigational agent or study drug within 30 days or 5 half-lives prior to Screening
* Receipt of any protein- or antibody-based therapeutic agent within 3 months prior to Screening
* Prior exposure to telotristat etiprate
* Use of tobacco, smoking cessation products, or nicotine products within 3 months prior to Screening
* History of major surgery within 6 months prior to Screening
* History of any GI surgery that may induce malabsorption
* History of renal disease, or significantly abnormal glomerular filtration rate (<90 mL/min as calculated using the Cockcroft-Gault equation) at Screening
* History of hepatic disease, or significantly abnormal liver function tests at Screening
* History of any clinically significant psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, endocrinologic, hematological, or GI abnormality
* History of any active infection within 14 days prior to Screening
* History of alcohol or substance abuse within 2 years prior to Screening
* Positive hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody) or positive human immunodeficiency virus antibody screens
* Concurrent conditions that could interfere with safety and/or tolerability measurements
* Donation or loss of >500 mL of blood or blood product within 3 months prior to Screening
* Women who are breastfeeding or are planning to become pregnant during the study
* Positive serum pregnancy test (females only)
* Positive urine screen for selected drugs of abuse and cotinine
* Consumption of alcohol within 48 hours prior to study start
* Consumption of caffeine- and/or xanthine-containing products within 72 hours of study start
* Consumption of grapefruit, Seville oranges, and grapefruit- or Seville orange-containing products within 72 hours prior to study start
* Unable or unwilling to communicate or cooperate with the Investigator for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of telotristat ethyl | Days 1, 2, 3, 6, 7, 8
Plasma concentration of metabolite LP-778902 | Days 1, 2, 3, 6, 7, 8

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Madison, Wisconsin, United States